CLINICAL TRIAL: NCT06234176
Title: Influence of Psychomotor Therapy on Quality of Life in Patients With a Major Depressive Disorder: a Randomized Controlled Trial
Brief Title: Impact of Psychomotor Therapy on the Quality of Life in Depression
Acronym: PsyMot-Dep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Principal Investigator, Aude Paquet, Psychomotor Therapist, Psychology PhD, Centre Hospitalier Esquirol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02678-37
Record Dates: First submitted 2024-01-15; First posted 2024-01-31 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: psychomotor therapy; quality of life; major depressive disorder; psychomotor profile; sensory processing
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Experimental Group: Personalised psychomotor therapy: 1 psychomotor therapy session of 45 minutes per week for 12 weeks + Duke Health Scale.
  The sessions will be based on static and dynamic body exercises involving muscle relaxation, breathing, sensations and moving the body.
  Control Group: Usual care for 12 weeks with a weekly telephone interview + Duke's Health Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised psychomotor therapy group (Experimental): 1 psychomotor therapy session of 45 minutes per week for 12 weeks + Duke Health Scale.
  Interventions: Behavioral: Personalised psychomotor therapy
- Usual treatment group (Active Comparator): Standard treatment for depression administered by a doctor + a weekly telephone interview for 12 weeks to administer the Duke Health Scale.
  Interventions: Other: Usual treatment

INTERVENTIONS:
Behavioral: Personalised psychomotor therapy — The content of the sessions will be personalised and determined solely by a qualified psychomotor therapist in charge of the patient, based on each participant's individual psychomotor profile, as determined from the initial assessment.
  The 12 sessions will take place with the same PT in a dedicated room at the centre where the patient is being treated. The sessions will consist of a range of playful static and dynamic body exercises, including exercises for emotional and tonic regulation, tonic-postural adaptation, and perceptual-motor adaptation.
  Not all participants in the GP group will have the same progression, nature or frequency of exercises over the 12 sessions.
  The study only allows for individual treatment. Other therapeutic approaches such as balneotherapy sessions, animal mediation, adapted physical activity programmes or targeted relaxation programmes are not permitted.
  During each session, the participant will be required to complete the Duke health profile.
  Other Names: GP
  Arms: Personalised psychomotor therapy group
Other: Usual treatment — Participants in the GC group will continue to receive their usual depression treatment without any changes to their prescribed therapies. Their participation in the study will involve weekly monitoring of their quality of life using the Duke scale. A nurse or psychomotor therapist will conduct this monitoring during a weekly fifteen-minute telephone interview. The follow-up will begin one week after the inclusion visit and will last for 12 weeks. Telephone appointments will be scheduled jointly with the participant based on their availability.
  Other Names: GC
  Arms: Usual treatment group

SUMMARY:
The effectiveness of psychomotor therapy in improving clinical outcomes or quality of life for individuals with depression is unclear.

The investigators will assess how the participants' quality of life and psychomotor profile change over time.

The study aims to compare the quality of life at 3 months between patients who received 3 months of personalised psychomotor therapy in addition to standard treatment and those who received standard treatment alone.

The study lasted for 6 months, and the investigators expects a total of 128 people to participate in this research across several hospital establishments. This study evaluates the effectiveness of two types of treatment, divided into two randomly selected groups.

To participate, individuals must have a medical diagnosis of major depressive disorder (MDD) and be between the ages of 20 and 60.

They must have depressive symptoms with an HDRS score greater than 16 and provide informed consent. They must be treated or hospitalised at the Centre Hospitalier Esquirol or the Centre Hospitalier Henri Laborit (France).

After providing consent, they will undergo an initial clinical interview that evaluates anxiety, self-esteem, pleasure, and quality of life. The therapist assessed the participant's muscle tone, gross motor skills, praxis, manual dexterity, rhythm, processing of sensory information, and body image.

Following the assessment, the participant was randomly assigned to either the experimental or control group.

The experimental group received the usual treatment for depression and underwent psychomotor therapy once a week for 12 weeks.

The control group received the standard treatment for depression and underwent weekly telephone interviews.

An assessment is scheduled at 1 month to evaluate the participant's health status, including any changes to treatment and assessment of anxiety and depressive symptoms.

Another interim check-up is scheduled at 3 months to assess the patient's health status. The interview will also assess any changes to treatment, anxiety and depressive symptoms, quality of life, and psychomotor function.

A final visit will be scheduled at 6 months for an assessment of the participant's health. The interview will also assess any changes to treatment, anxiety and depressive symptoms, quality of life, and psychomotor function.

DETAILED DESCRIPTION:
Hypothesis is that personalised weekly psychomotor therapy for 3 months (period of remission of depression) has a positive influence on the quality of life over time of people with MDD by improving their clinical (anxiety/anhedonia/psychomotor impairment) and psychomotor symptoms.

In this study, the investigators propose to compare the quality of life of two groups of participants: a group receiving one psychomotor therapy session per week in addition to the usual treatments for depression, and a group receiving the usual treatments for depression. The investigators will evaluate changes in quality of life and psychomotor profile over time (at 3 and 6 months).

Based on the results of our pilot study, the psychomotor examination will include an assessment of muscle tone, gross motor skills, praxis, manual dexterity, rhythm using the NP-MOT battery, sensory processing and body image.

Main objective To compare the quality of life at 3 months (M3) between MDD patients receiving 3 months of personalised psychomotor therapy in addition to standard treatment (GP) and those receiving standard treatment alone (GC).

Secondary objectives

1. To compare changes in quality of life over time between D0/M3, D0/M6 and M3/M6 in patients in the GP and GC groups; a difference between the groups will be sought.
2. Identify the psychomotor assessment items (tone, general motor skills, praxis, rhythm, body image, sensory profile) that differ at inclusion (D0) and 3 months (M3) between the GP and GC groups.
3. To identify clinical factors of depression (intensity of depression, anxiety, psychomotor slowing, anhedonia) associated with a difference in psychomotor profile at M3 between the GP and GC groups.
4. Identify items predictive of clinical improvement in depression based on psychomotor assessment items (tone, general motor skills, praxis, rhythm, body image, sensory profile) at 6 months (M6) in patients in the GP and GC groups.
5. Evaluate at M3, in the GP group, the number of sessions completed and the therapeutic alliance using a scale.

Primary outcome measure Difference at M3 between the GP and GC groups in the quality of life score assessed using the SF-36 (Short-Form 36 Health Survey) scale.

Secondary outcome measures

1. Difference between D0 and M3, D0 and M6, M3 and M6 in quality of life scores based on the SF-36.

   Change in Duke Health Profile scores over the 12 weeks of follow-up (S1 to S12).
2. Number and nature of assessment items that differ at inclusion and 3 months between GP and GC using the Neuropsychomotor Function Assessment Battery (NP-MOT), Body Image Questionnaire (BIQ), Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIAI-2), Adolescent/Adult Sensory Profile (AASP) tools
3. Depression intensity score on the Hamilton Depression Rating Scale (HDRS), anxiety intensity score on the Hamilton Anxiety Rating Scale (HARS), psychomotor slowing down score on the CORE scale, anhedonia score on the SHAPS scale, and body image score on the QIC and MAIA-2 scales, sensory profile scores on the AASP scale, frequency of tonic-emotional manifestations, sub-scores of the NP-MOT battery, at M3.
4. Clinical improvement score: 50% reduction in HDRS score, scores AASP, score QIC, score MAIA-2 and items sub-scores NP-MOT
5. Total number of sessions and score on the French version of the Therapeutic Alliance Session Rating Scale at M3

The inclusion criteria for participants in this study are as follows: being between the ages of 20 and 60, having a diagnosis of major depressive disorder according to DSM-5 criteria, having a HDRS score greater than 16 indicating major symptoms, and being hospitalized or receiving care at one of the participating centres.

Additionally, participants must be affiliated with or benefiting from a social security scheme.

The participant and investigator must sign a written consent form that is both free and informed. This must be completed no later than the day of inclusion and before any required research examinations.

Non-inclusion criteria for this study are: psychiatric co-morbidity (excluding tobacco addiction, eating disorders, bipolar disorder, obsessive-compulsive disorder, schizophrenia and related disorders), sensory disability or known neurological pathology, history of neurological damage to the brain (especially strokes, tumours, trauma resulting in loss of consciousness lasting more than 10 minutes), and limited functional ability (difficulty moving about, performing manual tasks or moving about).

Participants may be excluded from the study if they are unable to understand the questionnaires or related information, unable to travel to the inclusion centre via personal vehicle or public transport, pregnant or breastfeeding (as declared), subject to compulsory hospitalisation or under guardianship or trusteeship, or lack social protection.

The research is conducted as follows:

* Pre-selection by the coordinating investigator or co-investigator, validation of participation criteria by the referring doctor and information of participants by the referring doctor or coordinating investigator or staff associated with the research.
* Reflection period: between 24 and 72 hours.
* V0: Inclusion Collect of written consent, Socio-demographic data (age, sex, family situation, profession, place of residence, environment), psychiatric history, treatments received (medicinal and non-medicinal), etc.

Quality of life scale (SF36) Clinical assessments: Hamilton Depression Rating Scale (HDRS); Hamilton Anxiety Rating Scale (HARS); psychomotor slowing down scale (CORE), Rosenberg Self-Esteem Scale (EES-10), Anhedonia Scale (SHAPS) Psychomotor assessment: sensory profile (AASP), body image (QIC, MAIA-2), tone (NP-MOT); general motor skills (NP-MOT), rhythm (NP-MOT); praxis (NP-MOT); manual dexterity (PPT) Randomisation: allocation of patients by drawing lots to the GP (personalised psychomotor therapy in addition to standard treatment) or GC (standard treatment) groups.

GP: Personalised psychomotor therapy: 1 psychomotor therapy session of 45 minutes per week for 12 weeks + Duke Health Scale.

The sessions will be based on static and dynamic body exercises involving muscle relaxation, breathing, sensations and moving the body. For each session the Session Rating Scale will be use.

GC: Usual care for 3 months with a weekly telephone interview + Duke's Health Scale.

* V1: visit at 1 month ± 4 days for an interim assessment Treatments received and/or modified in the last 4 weeks Clinical assessments: HDRS; HARS; CORE, EES-10, SHAPS
* V2: visit at 3 months ± 7 days Treatments received and/or modified in the last 3 months Clinical assessments: HDRS; HARS; CORE, EES-10, SHAPS Number of psychomotricity sessions performed Quality of life scale (SF36) Blind psychomotor assessment: AASP, QIC, MAIA-2, NP-MOT
* V3: visit at 6 months ± 7 days Treatments received and/or modified in the last 3 months Clinical assessments: HDRS; HARS; CORE, EES-10, SHAPS Quality of life scale (SF36) Blind psychomotor assessment: AASP, QIC, MAIA-2, NP-MOT Participants in the GC group were offered 12 sessions of psychomotor therapy.

At V2, the psychomotor assessment will be carried out by a psychomotor therapist who has not provided psychomotor therapy to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depressive episode according to DSM-5 criteria.
* HDRS > 16
* Hospitalized or followed-up in one of the participating centers.
* Affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (no later than the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Psychiatric comorbidity (non-tobacco addiction, eating disorders, bipolar disorder, obsessive-compulsive disorder, schizophrenia and related disorders)
* Sensory impairment or proven neurological pathology
* History of neurological brain damage (including stroke, tumor, trauma resulting in loss of consciousness lasting more than 10 minutes)
* Limited functional ability (difficulty in moving about, performing manual tasks or moving about)
* Inability to understand questionnaires and study information
* Inability to travel to the inclusion center (personal vehicle, public transport)
* Pregnant or breast-feeding women, on declaration
* Forced hospitalization, subjects under guardianship or trusteeship, lack of social protection

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Difference in quality of life assessed using the Short-Form 36 Health Survey | at 3 month
  Difference between GP and GC groups in quality of life score

SECONDARY OUTCOMES:
Difference in time of quality of life using the Short-Form 36 Health Survey | first day to 6th month
  Difference between D0 and M3, D0 and M6, M3 and M6 in quality of life scores
Evolution of quality of life using the Duke health profile | first day to 6th month
  Evolution of Duke health profile scores from week 1 to week 12 in both GP and GC groups
Difference in psychomotor profile | 3th and 6 th month
  Number and nature of assessment items that differ at 1 and 3 months between GP and GC using NP-MOT, QIC, MAIA-2, AASP tools
Description of depression intensity using the Hamilton Depression Rating Scale | at 3 month
  clinical improvement concerning depression low score to Hamilton Depression Rating Scale indicate a low depressive intensity
Description of anxiety intensity using the Hamilton Anxiety Rating Scale | at 3 month
  clinical improvement concerning anxiety low score to Hamilton Anxiety Rating Scale indicate a low anxiety intensity
Description of psychomotor slowing using the CORE scale | at 3 month
  clinical improvement concerning psychomotor slowing low score to CORE Scale indicate a low psychomotor slowing
Description of anhedonia using the Snaith-Hamilton Pleasure Scale | at 3 month
  clinical improvement concerning anhedonia low score to Snaith-Hamilton Pleasure Scale indicate a low anhedonia intensity
Description of body image using the Multidimensional Assessment of Interoceptive Awareness | at 3 month
  clinical improvement concerning body image low score to Multidimensional Assessment of Interoceptive Awareness indicate a low interoceptive awarness
Description of sensory profile using the Adolescent Adult Sensory Profile | at 3 month
  clinical improvement concerning sensory profile The AASP is composed by four subscores
  * norm for low registration subcore is between 24-35
  * norm for sensation seeking subcore is between 43-56
  * norm for lsensory sensitivity subcore is between 26-41
  * norm for sensation avoiding subcore is between 27-41
Frequency of tonic-emotional manifestations | at 3 month
  observed reactions: awkward gestures, reassurance gestures, fixed smile, facial rictus, rigid body posture, contorting, stiffening, slightly theatrical posture, emotional uncontrol, neurovegetative manifestations: presence or absence
Frequency of psychomotor impairment using the NP-MOT battery | at 3 month
Frequency of sessions | at 3 month
  Therapeutic alliance is mesured by number of sessions completed by GP participants out of 12 planned sessions.
  Session Rating Scale scores for the 12 sessions completed by GP participants.

CONTACTS AND LOCATIONS:
Locations (1):
- CH Esquirol, Limoges, France